CLINICAL TRIAL: NCT00913159
Title: A Randomized Controlled Trial Comparing Efficacy of HM3 vs F2 Lithotripters for Stone Fragmentation
Brief Title: A Trial Comparing Efficacy of HM3 Versus F2 Lithotripters for Stone Fragmentation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Alana Desai, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alana Desai HM3 vs F2
Record Dates: First submitted 2009-06-01; First posted 2009-06-04 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Urolithiasis
Keywords: Renal stones; lithotripsy; stone free rate
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis | interventions — Lithotripsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Using HM3 lithotripter (Active Comparator): This is an older generation lithotripter
  Interventions: Procedure: Extracorporeal Shock Wave Lithotripsy (ESWL)
- F2 lithotripter (Active Comparator): This is a newer generation lithotripter
  Interventions: Procedure: Extracorporeal Shock Wave Lithotripsy (ESWL)

INTERVENTIONS:
Procedure: Extracorporeal Shock Wave Lithotripsy (ESWL) — Using electric shock wave to treat urolithiasis

SUMMARY:
The older lithotripter, HM3, has over 90% stone-free rate in most studies. However, it's less transportable than the new model, F2. There are no prospective trials performed to make a valid comparison between these 2 lithotripters in terms of efficacy of stone fragmentation and clinical outcomes.

DETAILED DESCRIPTION:
Shock wave kidney stone treatment was introduced in the 1980's. It is the least invasive method to treat kidney stone disease. The unmodified Dornier HM3 has over 90% stone free rate in most studies. The MH3 requires immersion in a full bath, necessitating dedicated operative space. The new generation model F2 uses water cushion as a coupling medium and is easily transported. The generators used in both machines are also different. The newer model has the advantage of being more convenient due to portability and ease of use of the coupling medium, but there have been no prospective studies to compare these 2 machines in terms of efficacy of stone fragmentation and clinical outcomes. We seek to compare the HM3 with the F2 models in terms of stone free rates, complications and clinical outcomes to determine which machine is the most effective and will limit the need for additional stone procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with urolithiasis and choose to have ESWL treatment
2. Age 18-90 years old
3. Able to understand the informed consent

Exclusion Criteria:

1. Minors
2. Cognitively impaired

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Stone free rate, complications and need for ancillary procedures | 3-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alana Desai, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Division of Urology, Washington University School of Medicine, St Louis, Missouri, United States